CLINICAL TRIAL: NCT03499067
Title: A Dispensing Clinical Trial of Invigor I Lens Against Clariti Lens
Brief Title: A Dispensing Clinical Trial of Test Contact Lens Against Marketed Contact Lens
Status: Completed | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-18-07
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to wear the test or control contact lens for 1 month and then crossed-over to wear the other contact lens for 1 month.
Who Masked: Participant, Investigator
Masking Description: This will be a double-masked study in which both participant and investigator will be masked.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Test lens (Experimental): Subjects wearing the test contact lens either as first or second pair during the cross-over study.
  Interventions: Device: Test lens; Device: Control lens
- Control lens (Active Comparator): Subjects wearing the control contact lens either as first or second pair during the cross-over study.
  Interventions: Device: Test lens; Device: Control lens

INTERVENTIONS:
Device: Test lens — Contact lens
  Other Names: Invigor I lens
Device: Control lens — Contact lens
  Other Names: Clariti lens

SUMMARY:
Evaluation of the clinical performance of an investigational silicone-hydrogel contact lens (test) compared to a marketed lens (control), when worn on a daily basis for 1 month.

DETAILED DESCRIPTION:
Evaluation of the clinical performance of an investigational silicone-hydrogel contact lens (test) compared to a marketed silicone- hydrogel contact lens (control), when worn on a daily basis for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Currently wears soft contact lenses.
* Requires spectacle lens powers between -0.75 to -6.50 diopters sphere (0.25D steps).
* Has no more than 0.75 diopters of refractive astigmatism.
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.
* Has a usable pair of spectacle lenses if required for transportation to the site for the initial visit

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.
* Known allergy to a product used in this study (ex. Shellfish allergy)
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research Center, University of California, Berkeley, Berkeley, California
  - Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens Then Control Lens: Subjects were randomized to wear test lens for one month then control lens for one month during the cross-over study.
  Test lens: Contact lens
  Control lens: Contact lens
- Control Lens Then Test Lens: Subjects were randomized to wear control lens for one month then test lens for one month during the cross-over study.
  Test lens: Contact lens
  Control lens: Contact lens
Period: First Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 27 | 31
Completed | 22 | 24
Not Completed | 5 | 7
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 3 | 6
Period: Second Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total participants
Arm/Group | Overall Study
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Lens Surface Wettability
Description: Lens surface wettability was measured on a scale of 0-4, 0.25 steps (0 Very Poor: Immediately displaying non-wetting areas on the lens surface, immediate drying time, 1 Poor: Irregular surface appearance, drying time << blink time, 2 Acceptable: Smooth surface appearance immediately, after the blink becoming irregular after a while, drying time ≤ blink time, 3 Good: Typical soft lens appearance with long drying time 4 Excellent: Appearance of a healthy cornea with very long drying time)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Lens: Subjects were randomized to wear test contact lens for one month in this cross-over study.
  Test lens: Contact lens
- Control Lens: Subjects were randomized to wear control contact lens for one month in this cross-over study.
  Control lens: Contact lens
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.26 (0.48) | 3.26 (0.44)

2. Primary Outcome: Lens Surface Wettability
Description: as for outcome 1
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.18 (0.53) | 3.25 (0.47)

3. Primary Outcome: Lens Surface Wettability
Description: as for outcome 1
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.11 (0.51) | 3.01 (0.62)

4. Primary Outcome: Lens Surface Deposits
Description: Lens surface deposits was measured on a Scale 0-4, 0.25 steps (0: Clean, no deposits, 1: 5 or less small deposits (<0.1mm), 2: >5 deposits of <0.1mm size or film covering 25-50% of surface, 3: Deposits of between 0.1 and 0.5mm or film covering 50-75% of surface, 4: Deposits of 0.5mm or larger or film covering more than 75% of surface)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.02 (0.12) | 0.04 (0.23)

5. Primary Outcome: Lens Surface Deposits
Description: Lens surface deposits was measured on a Scale 0-4, 0.25 steps (0: Clean, no deposits,1: 5 or less small deposits (<0.1mm), 2: >5 deposits of <0.1mm size or film covering 25-50% of surface, 3: Deposits of between 0.1 and 0.5mm or film covering 50-75% of surface, 4: Deposits of 0.5mm or larger or film covering more than 75% of surface).
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.30 (0.60) | 0.26 (0.53)

6. Primary Outcome: Lens Surface Deposits
Description: as for outcome 5
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.35 (0.54) | 0.38 (0.63)

7. Primary Outcome: Overall Lens Fit Acceptance
Description: Overall lens fit acceptance was measured on a scale of 0-4, 0.25 steps (0 Unacceptable-Can't be worn, 1 Acceptable -Poor/worn under supervision, 2 Acceptable -Fair, prefer refit, 3 Acceptable -Good, 4-Acceptable -Optimum)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.30 (0.33) | 3.27 (0.35)

8. Primary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 7
Time Frame: 2-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.28 (0.41) | 3.31 (0.35)

9. Primary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 7
Time Frame: 4-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 3.31 (0.36) | 3.13 (0.53)

10. Primary Outcome: Percentage of Participants With Optimum, Slightly Decentered, Extremely Decentered Lens Centration
Description: Lens Centration was assessed in primary gaze, white light, diffuse, 8xmag, with graticule on a grade of Optimum, Slightly decentered (<0.5mm), Extremely decentered (>0.5mm)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
percentage of participants
  Optimal | 49 | 38
  Slightly Decentered | 45 | 55
  Extremely Decentered | 6 | 7

11. Primary Outcome: Percentage of Participants With Optimum, Slightly Decentered, Extremely Decentered Lens Centration
Description: as for outcome 10
Time Frame: 2-weeks
Measure: Number; unit: percentage of participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
percentage of participants
  Optimal | 57 | 40
  Slightly Decentered | 43 | 52
  Extremely Decentered | 0 | 8

12. Primary Outcome: Percentage of Participants With Optimum, Slightly Decentered, Extremely Decentered Lens Centration
Description: as for outcome 10
Time Frame: 4-weeks
Measure: Number; unit: percentage of participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
percentage of participants
  Optimal | 59 | 33
  Slightly Decentered | 40 | 59
  Extremely Decentered | 1 | 8

13. Secondary Outcome: Bulbar Conjunctiva Hyperaemia
Description: Bulbar Conjunctiva Hyperaemia was measured on a scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 1.11 (0.49) | 1.11 (0.49)

14. Secondary Outcome: Bulbar Conjunctiva Hyperaemia
Description: Bulbar Conjunctiva Hyperaemia was measured on a scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 1.20 (0.45) | 1.23 (0.43)

15. Secondary Outcome: Bulbar Conjunctiva Hyperaemia
Description: Bulbar Conjunctiva Hyperaemia was measured on a scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 1.15 (0.47) | 1.27 (0.43)

16. Secondary Outcome: Limbal Conjunctiva Hyperaemia
Description: Limbal Conjunctiva Hyperaemia was measured on a Scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.57 (0.35) | 0.57 (0.35)

17. Secondary Outcome: Limbal Conjunctiva Hyperaemia
Description: Limbal Conjunctiva Hyperaemia was measured on a Scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.71 (0.40) | 0.63 (0.39)

18. Secondary Outcome: Limbal Conjunctiva Hyperaemia
Description: Limbal Conjunctiva Hyperaemia was measured on a Scale of 0-4, 0.25 steps (0=None, 4=Severe injection)
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 46 | 46
units on a scale | 0.65 (0.42) | 0.76 (0.35)

ADVERSE EVENTS:
Time Frame: From dispense up to 4-weeks on each type of lenses
Arm/Group | Test Lens | Control Lens
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03499067/Prot_SAP_000.pdf